CLINICAL TRIAL: NCT04134663
Title: Comparison of Direct and Indirect Effects of Intranasal Oxytocin Using Co-administration With a Vasoconstrictor
Brief Title: Comparison of Intranasal Oxytocin Effects Using Co-administration With a Vasoconstrictor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Keith Kendrick, Professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN-43
Record Dates: First submitted 2019-10-18; First posted 2019-10-22 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Healthy
Keywords: vasoconstrictor; oxytocin; EEG; peripheral nervous system response
MeSH Terms: interventions — Vasoconstrictor Agents

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- vasoconstrictor + intranasal oxytocin group (Experimental): subjects receive the vasoconstrictor followed by oxytocin
  Interventions: Drug: vasoconstrictor and oxytocin treatment
- vasoconstrictor's placebo + intranasal oxytocin group (Active Comparator): subjects receive the vasoconstrictor's placebo followed by oxytocin
  Interventions: Drug: vasoconstrictor's placebo and oxytocin treatment
- vasoconstrictor + intranasal oxytocin placebo group (Placebo Comparator): subjects receive the vasoconstrictor followed by intranasal oxytocin's placebo
  Interventions: Drug: vasoconstrictor and oxytocin's placebo treatment

INTERVENTIONS:
Drug: vasoconstrictor and oxytocin treatment — intransal administration of vasoconstrictor and oxytocin
  Arms: vasoconstrictor + intranasal oxytocin group
Drug: vasoconstrictor's placebo and oxytocin treatment — intransal administration of vasoconstrictor's placebo and oxytocin
  Arms: vasoconstrictor's placebo + intranasal oxytocin group
Drug: vasoconstrictor and oxytocin's placebo treatment — intransal administration of vasoconstrictor and oxytocin's placebo
  Arms: vasoconstrictor + intranasal oxytocin placebo group

SUMMARY:
This study aims to dissociate direct from indirectly mediated effects of intranasal oxytocin administration by using treatment with or without prior intranasal administration of a vasoconstrictor to reduce peripheral increases in peptide concentrations. Primary outcomes of the randomized placebo-controlled double-blind experiment are blood oxytocin concentration and oxytocin-associated responses in central and peripheral systems.

Intranasal application of the neuropeptide oxytocin has been reported to produce a number of neural, physiological and behavior effects which may be of potential therapeutic relevance, but it is unclear the extent to which they are mediated directly via the peptide entering the brain or indirectly as a result of increased peripheral concentrations. In the current placebo-controlled, double blind experiment on healthy adult male subjects the investigators will measure the effects of a single dose of intranasal oxytocin (24IU) on brain activity (using electroencephaolography - EEG) as well as on cardiac (heart-rate and heart-rate variablility) and gastric (electrogastrogram - EGG) activity and physiological arousal (skin conductance response - SCR). The pattern of functional effects observed will be compared with subjects receiving intranasal pretreatment with a vasoconstrictor prior to oxytocin in order to reduce the amount of oxytocin entering the peripheral circulation. The investigators hypothesize that prior administration of the vasoconstrictor will greatly reduce blood oxytocin concentrations following intranasal oxytocin treatment. Where neural/physiological effects are also affected, this will indicate an indirectly mediated action of intranasally administered oxytocin whereas if they are not this will indicate a directly mediated action.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects without past or current psychiatric or neurological disorders

Exclusion Criteria:

* history of head injury
* medical or psychiatric illness.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2019-03-02 (Actual); Primary Completion 2021-06-18 (Actual); Study Completion 2021-07-20 (Actual)

PRIMARY OUTCOMES:
blood oxytocin concentration | 2 hours
  blood oxytocin concentration changes following vasoconstrictor/placebo and oxytocin/placebo treament
resting EEG time-frequency | 2 hours
  resting EEG time-frequency changes following vasoconstrictor/placebo and oxytocin/placebo treament

SECONDARY OUTCOMES:
heartrate | 2 hours
  heartrate (and heartrate variability) changes following vasoconstrictor/placebo and oxytocin/placebo treament
skin conductance | 2 hours
  skin conductance level (measured by skin conductance response) changes following vasoconstrictor/placebo and oxytocin/placebo treament
gastrointestinal activity | 2 hours
  gastrointestinal activity (measured by electrogastrogram) changes following vasoconstrictor/placebo and oxytocin/placebo treament

CONTACTS AND LOCATIONS:
Locations (1):
- school of life science and technology, University of Electronic Science and Technology of China, Chengdu, Sichuan, China